CLINICAL TRIAL: NCT02099474
Title: Evaluation of the Pharmacokinetic Properties and the Tolerance of Raltegravir During the Third Trimester of Pregnancy
Brief Title: Evaluation of Raltegravir During the Third Trimester of Pregnancy
Acronym: ANRS 160 RalFE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 160 RalFE; 2013-004571-12 (EudraCT Number)
Record Dates: First submitted 2014-03-19; First posted 2014-03-31 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: HIV-1 Infection; PREGNANCY
Keywords: HIV-1; HIV mother to child prevention; Raltegravir; Pharmacokinetic
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltegravir (Experimental): All women have been prescribed raltegravir before study participation.
  Interventions: Other: Study of pharmacokinetic properties of raltegravir during the 3rd trimester of pregnancy

INTERVENTIONS:
Other: Study of pharmacokinetic properties of raltegravir during the 3rd trimester of pregnancy — Introduction of a catheter for performing 5 blood samples in pregnant women infected by HIV-1, before the raltegravir intake, 0.5, 3, 8 and 12 hours after the intake at each of two visits (between 30 and 37 weeks of amenorrhea, and 4 to 6 weeks after delivery)
  Other Names: raltegravir (Isentress®)

SUMMARY:
The purpose of this study is to assess the evolution of raltegravir concentration in the mother (between the 3rd trimester of pregnancy and one month post-delivery) and her neonate, when this drug is used to prevent mother-to-child HIV-1 transmission as part of a combined antiretroviral regimen.

DETAILED DESCRIPTION:
1. Objectives

   1. Principal objective

      * To study pharmacokinetic properties of raltegravir in pregnant women infected by HIV-1, during the third trimester of pregnancy (between 30 and 37 weeks of amenorrhea) and 1 month after childbirth (between W4 and W6 postpartum), as well as in their neonate.
   2. Secondary objectives

      * Estimate the frequency of women receiving raltegravir and having indetectable viral load at delivery (and those having a strictly indetectable viral load, with no signal under the threshold of the technique used).
      * Describe the tolerance to raltegravir in pregnant women during the third trimester and in her neonates
2. Methodology

   * National multicenter pharmacokinetic study conducted among pregnant women infected by HIV-1 and exposed to raltegravir during pregnancy.
3. Statistical method

   * Method of population pharmacokinetic with 5 samples: before the drug intake, 0.5, 3, 8 and 12 hours after the intake at each of the 2 visits (between 30 and 37 weeks of amenorrhea, and 4 to 6 weeks after delivery).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman, between 30 and 37 weeks of amenorrhea
* 18 years old and over
* Infected by HIV-1
* Receiving a therapeutic combination, stable for at least 15 days before inclusion, with raltegravir at the standard dose (400 mg twice daily) which the doctor plans to maintain till the end of pregnancy and at least one month after delivery
* Informed consent signed by mother and investigator (at the latest day of pre-inclusion and before any examination conducted as part of research)
* Affiliated person or beneficiary of a social security system (medical aid of state or AME is not a social security system)
* Participant agreeing to be registered in the national file of the people who participate in biomedical researches

Exclusion Criteria:

* Infected by HIV-2
* Under 18 years old
* Receiving therapeutic association with atazanavir (Reyataz®), fosamprenavir (Telzir®), or efavirenz ( contained in Sustiva® and Atripla®)
* Currently using medication, drugs or alcohol which can interfere with the research: rifampicine, phénobarbital, phénytoïne, topical gastrointestinal, antiacid and adsorbents
* Presenting a clinical situation or acute pathology incompatible with the realisation of a pharmacokinetic study.
* Planned absence which could hinder research participation (travel abroad, moving, imminent transfer ...)
* Participating in another research, except the French perinatal survey (ANRS CO1 EPF or ANRS CO11 observatory), including an exclusion period still in progress at the pre-inclusion
* Person under guardianship, or deprived of freedom by a judicial or administrative decision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the AUC and raltegravir trough concentration during and after pregnancy | 5 samples: before the drug intake, 0.5, 3, 8 and 12 hours after the intake at each of the 2 visits (between 30 and 37 weeks of amenorrhea, and 4 to 6 weeks after delivery)

SECONDARY OUTCOMES:
Estimation of placental transfer of raltegravir | Up to 72 hours after delivery
  Cmin, Cmax, AUC, t1/2 of raltegravir in newborns.
Study of genetic polymorphism which could modify raltegravir concentrations | Up to 72 hours after delivery
Proportion of women having a viral load < 50 cp/mL at delivery | Up to 72 hours after delivery
Proportion of maternal-to-child HIV transmission | Up to 72 hours after delivery
Untimely stop of raltegravir for toxicity or intolerance | Up to 72 hours after delivery
Clinical and biological anomaly occurring during the third trimester of pregnancy and during the first 6 months of life of the neonate. | Month 6
  Number of newborns with adverse events as a measure of safety and tolerability. Newborns will be followed up to 24 weeks of age.
Estimation of neonatal elimination of raltegravir | Up to 72 hours after delivery
  Cmin, Cmax, AUC, t1/2 of raltegravir in newborns.

CONTACTS AND LOCATIONS:
Overall Officials: JADE GHOSN, MD, Principal Investigator — CHU Hôtel Dieu PARIS
Locations (1):
- CHU Hôtel Dieu, Paris, France

REFERENCES:
- [Derived] Zheng Y, Hirt D, Delmas S, Lui G, Benaboud S, Lechedanec J, Treluyer JM, Chenevier-Gobeaux C, Arezes E, Gelley A, Amri I, Urien S, Bouazza N, Foissac F, Warszawski J, Ghosn J. Effect of Pregnancy on Unbound Raltegravir Concentrations in the ANRS 160 RalFe Trial. Antimicrob Agents Chemother. 2020 Sep 21;64(10):e00759-20. doi: 10.1128/AAC.00759-20. Print 2020 Sep 21. PMID 32661003